CLINICAL TRIAL: NCT00214318
Title: The Effects of ß2 Polymorphisms on Beta Selectivity After ß-adrenergic Blockade in Patients With Heart Failure
Brief Title: Beta-2 Polymorphisms and Beta Receptor Selectivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-2005-0006
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Terbutaline; Metoprolol; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Terbutaline plus Metoprolol or carvedilol

SUMMARY:
We hypothesize that b2 adrenergic polymorphisms affect b-receptor selectivity in patients with heart failure treated with either a b1-selective or a b-nonselective agent. b-2 polymorphisms may contribute to differing responses to drug treatment with beta-blockers in heart failure. Characterizing these polymorphisms may help explain the variability in the degree of "selectivity" of action of b-blockers at the b receptor, namely if their action is specific for the b-1 or b-2 receptor. Part A was conducted at the University of Utah, and all subjects completed study related activities. Part B (sub-study) consists of genotyping of blood samples collected in part A, which will be completed at the University of Wisconsin. Sub-study (samples and DNA isolation) or Part B entailed analyzing an extra 10 mL of blood that was taken for DNA isolation. Genotyping (i.e. determination of genetic makeup) of beta adrenergic polymorphisms utilized polymerase chain reaction followed by pyrosequencing.

ELIGIBILITY:
Inclusion Criteria:

* systolic dysfunction with ejection fraction ≤40%
* symptomatic heart failure class 2-3
* >18 years of age
* optimal medical therapy of HF excluding the use of any beta-blockers within the previous 30 days of the study

Exclusion Criteria:

* active myocarditis
* hemodynamically significant valvular heart disease
* hypertrophic cardiomyopathy
* contra-indications to beta-blockers
* concomitant use of beta-agonists
* beta-antagonist or anti-arrhythmics
* unstable angina
* myocardial infarction or bypass surgery within 3 months
* significant renal insufficiency [creatinine >2.5 mg/dL], liver disease, or anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-01; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The effect of beta-2 polymorphisms on potassium changes in response to terbutaline infusions

CONTACTS AND LOCATIONS:
Overall Officials: orly vardeny, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States